CLINICAL TRIAL: NCT00730964
Title: A Post-marketing Surveillance Study of the Occurrence of Serious Adverse Reactions Among Patients Who Receive Optison in Routine Medical Practice
Brief Title: A Prospective Surveillance Trial to Evaluate the Safety of Optison in Clinical Practice.
Acronym: OSSAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GE-191-003
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-05

CONDITIONS: Echocardiography
Keywords: Surveillance; Optison; Perflutren; Echocardiography; Subjects receive Optison during enhanced echocardiography
MeSH Terms: interventions — FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 4 (Other): Open Label
  Interventions: Drug: Perflutren Protein-Type A Microspheres Injectable Suspension, United States Pharmacopeia (USP)

INTERVENTIONS:
Drug: Perflutren Protein-Type A Microspheres Injectable Suspension, United States Pharmacopeia (USP) — The recommended dose of Optison is 0.5mL injected into a peripheral vein. This may be repeated for further contrast enhancement as needed.
  The injection rate should not exceed 1mL per second. Follow the Optison injection with a flush of 0.9% sodium chloride injection, USP or 5% dextrose in water injection, United States Pharmacopeia (USP) .
  The maximum total dose should not exceed 5.0mL in any 10 minutes period. The maximum total dose should not exceed 8.7mL in any one patient study.
  Other Names: Optison

SUMMARY:
This prospective surveillance trial will gather safety information for Optison when it is used in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* The subject is over 18 years old.
* The subject has been scheduled for an Optison-enhanced echocardiography exam.
* The subject has provided signed and dated informed consent.

Exclusion Criteria:

* Known hypersensitivity to perflutren, blood, blood products or albumin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1039 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Sheng, MD, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Optison: Open Label with 1039 subjects that received Optison to evaluate the safety of the product
Period: Overall Study
Arm/Group | Arm 1 - Optison
Started | 1039
Completed | 1039
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 - Optison
Number analyzed (Participants) | 1039
Age Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.99)
Age, Customized [Number; unit: participants]
  <=65 years | 671
  Between 65 and 75 years | 227
  >=75 years | 141
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 391
  Male | 648
Region of Enrollment [Number; unit: participants]
  United States | 1039

OUTCOME MEASURES:

1. Primary Outcome: The Frequency of Serious Adverse Reactions (SAR)'s Among Subjects Who Receive Optison (Causally Related to the Product)During Contrast Enhanced Echocardiography in Routine Clinical Practice.
Description: A Serious Adverse Reaction or (SAR) is considered causally related to the Optison product administered by the investigator. This reaction, should it occur, will be counted as a serious adverse reaction.
Time Frame: Within 24 hours post contrast administration
Measure: Number; unit: Serious Adverse Reactions
Arm/Group | Arm 1 - Optison
Number analyzed (Participants) | 1039
Serious Adverse Reactions | 0

2. Secondary Outcome: The Frequency of Overall Serious Adverse Events (SAE's) Among Subjects Who Receive Optison (Whether Related to the Product or Not) During Contrast Enhanced Echocardiography in Routine Clinical Practice.
Description: The frequency of any serious adverse event (SAE) whether it is related to the Optison product or not, after the administration of the Optison product during contrast enhanced echocardiography.
Time Frame: Within 24 hours post contrast administration
Measure: Number; unit: Serious adverse events
Arm/Group | Arm 1 - Optison
Number analyzed (Participants) | 1039
Serious adverse events | 6

ADVERSE EVENTS:
Arm/Group | Arm 1 - Optison
Serious Adverse Events (participants affected / at risk) | 5/1039
Other Adverse Events (participants affected / at risk) | 69/1039
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Optison (N=1039)
Non-sustained ventricular tachycardia (Cardiac disorders) | 1 (1)
Left Ventricular thrombus (Cardiac disorders) | 1 (1)
Fluid Overload (Vascular disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Left Ventricular Mass Requiring Surgery (Cardiac disorders) | 1 (1)
Episodes of Sustained Ventricular Tachycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Optison (N=1039)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 69 (288)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No